CLINICAL TRIAL: NCT04017481
Title: Development and Clinical Validation of a Rehabilitation Platform Based on Neuromodulation for Patients With Motor Control Disorders
Brief Title: Non Invasive Neuromodulation for Patients With Motor Control Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Collaborators: National Research Council, Spain (Other Government); Hospital Beata María Ana (Other); Hospital Universitario de Fuenlabrada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NeuroMOD
Record Dates: First submitted 2019-07-02; First posted 2019-07-12 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2019-07

CONDITIONS: Parkinson Disease
Keywords: neuromodulation; TMS; NFB
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Each study participant is assigned to one of the arms. Four intervention groups are defined as rTMS only, NFB only, both TMS and NFB, or neither TMS or NFB
Who Masked: Outcomes Assessor
Masking Description: Final outcomes evaluators are blinded. Clinical evaluation is performed using videotaped neurological examination. Neurophysiological evaluation is done with the raw data recorded during the sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Repetitive stimulating transcranial stimulation (rTMS) (Experimental): Subjects receive 8 sessions M1 Neuromodulation using rTMS according to the protocol ( 80% resting motor threshold, 10 Hertz; 1000 pulses; 25 trains de 4 seconds con 25 seconds intertrain.
  Interventions: Other: Repetitive transcranial magnetic stimulation (rTMS)
- EEG guided Neurofeedback (NFB) (Experimental): Subjects receive 8 sessions M1 EEG guided NFB with virtual reality goggles in order to modify the beta rhythm. The sessions have a duration of 20min
  Interventions: Other: EEG guided Neurofeedback (NFB)
- rTMS + NFB (Experimental): Subjects receive both interventions sequentially
  Interventions: Other: Repetitive transcranial magnetic stimulation (rTMS); Other: EEG guided Neurofeedback (NFB)
- No intervention (No Intervention): No interventions, the patient just comes to be evaluated sequentially according to the timing of experimental groups.

INTERVENTIONS:
Other: Repetitive transcranial magnetic stimulation (rTMS) — The intervention intends to change the cortical plasticity in specific cortical areas. rTMS is a non-invasive exogenous neuromodulation technique that uses repetitive magnetic pulses administered in a specific area of the head in order to influence the connectivity of the underlying brain area.
  Arms: Repetitive stimulating transcranial stimulation (rTMS); rTMS + NFB
Other: EEG guided Neurofeedback (NFB) — The intervention intends to change the cortical plasticity in specific cortical areas. The NFB is a non-invasive endogenous technique that seeks the self-regulation of cortical activity through the information represented in a videogame which is used to interact with the subject.
  Arms: EEG guided Neurofeedback (NFB); rTMS + NFB

SUMMARY:
Movement disorders are neurological syndromes leading to excessive movements or to limited control of voluntary and automatic movements. Many of these disorders are not life-threatening but represent serious difficulties in carrying out the activities of daily living and reduce patient's independence and quality of life.

This project NeuroMOD (neuromodulation for patients with disorders of motor control) proposes the development of a neuromodulation-based platform for the rehabilitation and restoration of motor and cognitive functions of patients suffering from Parkinson's disease (PD). Our project will focus on the application of a novel neurorehabilitation strategy, its functional and clinical validation, and on the evaluation of the impact of the use of the technologies involved in the musculoskeletal and the nervous system as well as user behavior.

Parkinson's disease was selected as target pathology since it represents a paradigm of motor disorder diseases.

Parkinson's disease affects adults and has a very high prevalence and a very high functional impact.

In order to achieve this objective, we have defined the following research areas:

Subproject 1. NeuroMOD: development of a neuromodulation platform composed by a TMS system, and an EMG (electromyography) and EEG (electroencephalography) system in combination with a system of virtual reality based on immersive glasses.

Subproject 2. NeuroMOD-PD: development of therapies and evaluation of clinical evidence and motor and cognitive impact of NeuroMOD in the rehabilitation of patients suffering from Parkinson's disease impact.

Subproject 3. NeuroMOD-Image: development of neuroimaging techniques to investigate the brain areas affected by the proposed therapies and temporary terms that neural plasticity is induced and evolves in Parkinson´s Disease.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinsons Disease
* Hoehn Yahr Scale I-III
* No drug changes in the last 90 days
* No exclusion criteria

Exclusion Criteria:

* Dementia (Minimental scale score <25)
* Dependency (modified Rankin scale > 3)
* Pregnancy or pregnancy plans
* Pacemaker
* Implanted metal devices
* cochlear implants
* claustrophobia
* drug infusion pumps
* epilepsy / epileptiform anomalies in electroencephalography (EEG)
* known structural alterations in magnetic resonance imaging (MRI)
* Atypical Parkinsonism
* Previous repetitive transcranial magnetic stimulation (rTMS)
* Severe comorbidity (cancer, severe debilitating diseases, etc.)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Motor changes | The day before the first stimulation session and 2 weeks after the first stimulation session
  UNIFIED PARKINSON'S DISEASE RATING SCALE (UPDRS) part III ( total values from 0-68, higher score worse clinical situation)
Motor changes | t2(2 weeks after finishing the protocol)
  UNIFIED PARKINSON'S DISEASE RATING SCALE (UPDRS) part III ( total values from 0-68, higher score worse clinical situation)
Neurophysiological cortical changes | The day before the first stimulation session and 2 weeks after the first stimulation session
  Cortical silent period measured using transcranial magnetic pulse in M1 and simultaneous register of electromyographical response
Neurophysiological cortical changes | t2(2 weeks after finishing the protocol)
  Cortical silent period measured using transcranial magnetic pulse in M1 and simultaneous register of electromyographical response

SECONDARY OUTCOMES:
Quality of life changes | t2(2 weeks after finishing the protocol)
  Changes in PDQ 39 (The 39-Item Parkinson's Disease Questionnaire) score, common range of 0-100 (100 = maximum level of problems).
Encephalographic changes | t2(2 weeks after finishing the protocol)
  Changes in microstates of electro encephalography (presence of state A, B, C, D and E)
Cognitive changes in objective measures of processing speed | t2(2 weeks after finishing the protocol)
  Changes in cognitive processing speed using computer based reaction time task

CONTACTS AND LOCATIONS:
Overall Officials: Juan Pablo Romero Muñoz, MD PhD, Principal Investigator — Universidad Francisco de Vitoria, Facultad de Ciencias Experimentales

IPD SHARING:
Plan to Share IPD: Yes
Individual anonymized participant data will be available to other researchers under request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: six months after the end of the study
Access Criteria: Individual anonymized participant data will be available to other researchers under request.

REFERENCES:
- [Derived] Romero JP, Moreno-Verdu M, Arroyo-Ferrer A, Serrano JI, Herreros-Rodriguez J, Garcia-Caldentey J, Rocon de Lima E, Del Castillo MD. Clinical and neurophysiological effects of bilateral repetitive transcranial magnetic stimulation and EEG-guided neurofeedback in Parkinson's disease: a randomized, four-arm controlled trial. J Neuroeng Rehabil. 2024 Aug 5;21(1):135. doi: 10.1186/s12984-024-01427-5. PMID 39103947